CLINICAL TRIAL: NCT02603133
Title: Web-based Implementation for the Science of Enhancing Resilience Study
Acronym: WISER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Duke University (Other)
Responsible Party: Principal Investigator, Jochen Profit, Associate Professor of Pediatrics, Director of Perinatal Health Systems Research, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-34547; R01HD084679 (NIH)
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Burnout, Professional; Resilience, Psychological
Keywords: healthcare; burnout; resilience; fatigue; NICU; safety culture; quality of care
MeSH Terms: conditions — Burnout, Professional; Burnout, Psychological; Fatigue

STUDY DESIGN:
Intervention Model Description: Participants are individually randomized to one of two cohorts. 1 cohort will serve as the waitlist control for Cohort 1 before starting their version of the intervention. Each cohort will experience slightly different versions of WISER, which only differ by the spacing of the intervention. Cohort 1 will receive a 10-day sequential (Seq) and a 10-day non-sequential (NSeq) rollout of the resilience tools. Seq will receive the tools on ten consecutive days. NSeq will receive messages daily with the exception of Thursdays, Fridays and Saturdays. Our tracking of attrition in the first study showed marked declines in participation on Thursdays, Fridays, and to some extent on Saturdays, but an increase on Sundays, hence this design to test a new way of counteracting attrition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Other): The intervention will begin for all NICUs, with baseline surveys as necessary pre-work. For those unable to attend, a link to the baseline survey will be emailed with site champion instructions to complete in groups at staff meetings and during shift change. Two weeks later, three randomly (random number generator) assigned NICUs (block 1) included in the first block webinar will then receive Module 1 of the intervention with Modules 2-6 being rolled out monthly. The second block of three NICUs starts approximately six-month later.
  Interventions: Behavioral: Three Good Things; Behavioral: Gratitude; Behavioral: Random Acts of Kindess; Behavioral: Awe; Behavioral: 1 Good Chat
- Cohort 2 (Other): This second block of 3 NICUs will start approximately six-months after roll-out of group 1. At time point 0 this NICUs in this group will receive a lecture on safety culture, unrelated to the burnout intervention.
  Interventions: Behavioral: Three Good Things; Behavioral: Gratitude; Behavioral: Random Acts of Kindess; Behavioral: Awe; Behavioral: 1 Good Chat
- Cohort 3 (July cohort) WISER 2.0 (Experimental): Individually randomized to one of two cohorts. Cohort 1 to start will serve as the waitlist control 1 before starting their version of the intervention. Each cohort will experience modified versions of WISER, which only differ by the spacing of intervention. Participants will receive 10-day sequential or 10-day non-sequential rollout of the resilience tools. Seq will receive the tools on ten consecutive days. NSeq will receive messages daily noThursdays, Fridays and Saturdays.
  Days 1 through 3 will be offered 3GT. Day 4 will continue with 3GT but add a single day activity for Gratitude. Day 5 adds a single activity for Awe. Day 6 adds a single day activity for RAK. Days 7 -10 the participant is offered the choice of Gratitude, Awe or RAK to accompany their daily 3GT. At 1 month follow-up time point, participants will receive 8 days of the 1 Good Chat tool, as a booster. At 6 month follow-up, participants will receive a gratitude exercise.
  Interventions: Behavioral: Three Good Things; Behavioral: Gratitude; Behavioral: Random Acts of Kindess; Behavioral: Awe; Behavioral: 1 Good Chat

INTERVENTIONS:
Behavioral: Three Good Things — In this tool participants reflect on "good things" that happened that day during evenings across 10 days. Participants are also able to voluntarily share their good things and read other participants' good things through the nightly anonymous log. By savoring good moments from earlier that day, participants are thought to shift from the natural focus on "what went poorly" due to negativity bias1 to an appreciation for what went well. This shift in focus is thought to reduce rumination and depression symptoms. In prior research, 3GTs was found to increase happiness and decrease depression in internet participants.2 In prior cohorts of 3GTs, we saw improvements in burnout, depression symptoms, work-life balance, and happiness. Participants also report benefiting from viewing nightly Three Good Things logs of others.
  Other Names: 3GT Tool
Behavioral: Gratitude — In this tool participants are offered the opportunity to cultivate gratitude toward others through a guided gratitude letter writing exercise.2 Through expressing gratitude, we learn more about our vital connections to others, often in surprising and meaningful ways. Previous research has found that gratitude interventions increase well-being in a number of ways, particularly in boosting positive affect.
  Other Names: Grat Tool
Behavioral: Random Acts of Kindess — In this tool, participants report kind acts that they have committed, received, and/or witnessed, each day. By committing random acts of kindness participants experience a boost of positive emotions, and report lower negative affect. Recipients of acts of kindness benefit as well.
  Other Names: RAK Tool
Behavioral: Awe — This tool provides participants the opportunity to recount in detail one of their own experiences of awe, and encourages them to be on the lookout for new ones (even minor examples) over a few days. When we experience awe, our sense of time expands, we are kinder to others, we experience higher life satisfaction, and we prefer experiences over material things.
  Other Names: Awe Tool
Behavioral: 1 Good Chat — This tool uses the latest research on cultivating relationships and increasing social connection. Feeling socially connected is linked to health and well-being outcomes, including longevity.6 The 1 Good Chat tool asks participants to reflect on good conversations and to note the prosocial behaviors that he/she and the other person engaged in
  Other Names: Good Chat Tool

SUMMARY:
Resilience means a healthcare provider's ability to cope, recover, and learn from stressful events, as well as their access to resources that promote health and well-being. Neonatal intensive care unit (NICU) health professionals' need to have particularly good resilience, because their work is extremely stressful and their patients, fragile preterm infants, require their undivided attention. The investigators propose a feasible and engaging intervention to enhance resilience among NICU health professionals promoting their ability to provide safe care.

DETAILED DESCRIPTION:
Optimizing provider well-being is critical to the delivery of safe and high quality care to the most vulnerable of patients: very preterm babies.

Major innovative objectives of this proposal include testing the Web-based Implementation for the Science of Enhancing Resilience (WISER) program's effectiveness in enhancing resilience among Neonatal Intensive Care Unit (NICU) health workers, evaluating its effect on unit safety culture, and examining its effect on clinical outcomes in preterm infants. The WISER program is an established but low-intensity yet engaging intervention, which integrates education and behavior modification to boost provider well-being and resilience in order to create an organizational environment which prevents patient harm.

Care for the more than 50,000 very low birth weight (VLBW; < 1500 gm) infants born annually in the United States is challenging and expensive. Quality of care and outcomes vary widely. Increasing technical demands and patient acuity have pushed burnout among health workers to the breaking point. The few tested interventions that improve caregiver resilience lack feasibility for widespread adoption. This study is designed to achieve the following aims:

1. Test the effectiveness of WISER in improving NICU health professional resilience;
2. Test the effectiveness of WISER in improving patient safety and organizational outcomes;
3. Test the sustainability of WISER; and
4. Describe the barriers and facilitators of the WISER program.

The investigators will test the efficacy of the WISER Program in the NICU setting using a stepped-wedge mixed-methods randomized controlled trial (swRCT) at six tertiary care NICUs. The results of this trial will also provide insights into the causal relations between health worker resilience, the organizational environment, and clinical outcomes among infants born VLBW.

Two blocks with 3 NICUs each will be randomly assigned to one of two intervention cohorts. The WISER NICUs program consists of six 10-minute videos delivered over the course of a six-month period. Following the end of the initial intervention, each NICU will receive individualized feedback/refresher webinar at 12 months, and a final follow-up at 24 months. The investigators will use measures of perception (surveys of health professional's perceptions) and quantifiable measures (clinical measures) to assess the efficacy of the intervention in different domains (resilience, organizational environment, and health). Qualitative methods will provide further insights into facilitators and barriers of the efficacy of WISER.

ELIGIBILITY:
Inclusion Criteria:

1. Location: newborn center, i.e. the NICU or a step down unit
2. Provider:

   1. Primary work place is the Newborn Center
   2. Full time equivalent of >=40%
   3. Date of hire more than 4 weeks prior to start of the intervention
3. Provider groups:

   1. Attendings that identify your newborn center as their primary site of work (not physicians from satellite NICUs)
   2. NICU fellows
   3. Nurse practitioners
   4. Physician Assistants
   5. Nurses, including nurse leadership (managers, educators)
   6. Nurse Assistant
   7. Respiratory care providers
   8. Transport specialists if primarily neonatal transport team
   9. Newborn Center Social workers
   10. Newborn Center Clerks
   11. Newborn Center Pharmacists
   12. Newborn Center Physical, Occupational, Speech, and Developmental Therapists
   13. Newborn Center Nutritionists
   14. Newborn Center Lactation Consultants

Exclusion Criteria:

1. Location: Labor and delivery or the newborn nursery
2. Provider: Work is delivered mostly outside the newborn center (this may affect providers who delivery services across the hospital such as residents, surgeons, anesthesia, consultants, nutritionists, PT/OT (these are included if they are mostly dedicated to the newborn center)
3. Float personnel
4. Does not speak english
5. Cannot operate computer or smart phone

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2650 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
NICU health professional resilience | 10 days, 1 month, 6 months, 12 months
  Burnout (emotional exhaustion) is the primary resilience outcome. The Maslach Burnout Inventory (MBI) has been the gold standard tool in the field of burnout research. In our investigations, the Emotional Exhaustion subscale, in particular, is consistently associated with variables such as staff turnover, disruptive behavior, productivity, delays, and teamwork. When used as a "percent agree" metric, we have shown it to be a very effective indicator of emotional exhaustion at the group level for a clinical area or work setting. We will use a shortened 4-item version of this subscale from the Maslach Burnout Inventory, which we validated in the NICU setting. The response scale ranges from 1 (disagree strongly) to 5 (agree strongly). Resilience will be calculated as the percentage of NICU providers who disagree slightly or strongly with the 4 items assessing features of emotional exhaustion.

SECONDARY OUTCOMES:
Work-Life Balance | 10 days, 1 month, 6 months, 12 months
  Work-Life Balance (WLB). WLB items were adopted from the College Activities and Behavior Questionnaire. These items that can be interpreted at face-value. All items are prefaced with, "during the past week, how often did this occur" and include items such as "argued with a co-professional" and "arrived home late from work"; they are answered on a four-point scale (0 = rarely or none; 3 = all of the time). Each of these items individually is face-valid and interpretable, but together they make for robust debriefings and discussions linking QI to work-life balance. They are internally consistent, with a Cronbach's alpha of α = 0.82 in our large resilience database.
Depressive symptoms | 10 days, 1 month, 6 months, 12 months
  The Center for Epidemiological Studies Depression Scale-10-item version (CES-D10), a psychometrically sound tool for screening respondents for clinical depression, consists of ten items. All items are prefaced with, "during the past week, how often did this occur," include items such as "I could not 'get going'" and "my sleep was restless," and are answered on a four-point scale (0 = rarely or none; 3 = all of the time). Each participant's responses are summed together to achieve a 0- to 30-point scale. A score of 10 or higher is considered a positive screen. We have used the CES-D10 in several WISER and three good things studies without any problems under the existing IRB. The CES-D10 is not a suicide screening tool, it is explicitly used to screen for depression without a suicide item.
Happiness | 10 days, 1 month, 6 months, 12 months
  Rather than to solely focus on negative outcomes, we will also measure happiness via the well-validated Subjective Happiness Scale. This 4-item measure of global subjective happiness was developed and validated 15 years ago using 14 studies with a total of 2732 participants, and has high internal consistency, test-retest, self-peer correlations, as well as excellent convergent and discriminant validity. The strong psychometrics and brevity of this scale have made it very popular in positive psychology interventions that require more precision in the assessment of subjective happiness.

OTHER OUTCOMES:
Safety and teamwork climate | 6 months and 12 months
  These two scales of the Safety Attitudes Questionnaire (SAQ) to assess health professionals' perceptions of these dimensions. Response scales range from 1 (disagree strongly) to 5 (agree strongly). These scales have been linked most closely with burnout, clinical, and operational outcomes. Scale scores will be calculated according to published methods.
Clinical delays in patient care | 6 month, 12 months
  All participants will receive a question on the survey regarding clinical delays in patient care. The response scale matches the SAQ.
Any health care associated infection | 12 months
  We will use standardized Vermont Oxford Network (VON) data definitions for all clinical data during the birth hospitalization. We chose this outcome because we have found it to be modifiable, and sensitive to health professional participation and unit safety culture. The VON addresses measurement bias through data collection procedures designed to minimize error and maximize accuracy. Data are abstracted from the medical record locally, using standardized protocols. Throughout this study, we will be able to collect routine clinical data collected for the VON database directly from participating NICUs.
Voluntary Nursing Turnover | 12 months
  This measure will be collected through a 3-item intention to leave index (I would like to find a better job; I often think about leaving this job; and I have plans to leave this job within the next year (α=.915)). We have found these items responsive to intervention in our work with the Comprehensive Unit Based Safety Program.
Conflicts with co-professionals | 6 months, 12 months
  Conflicts will be measured using a disruptive behavior index that assesses the prevalence of 15 distinct types of disruptive behaviors, as well as the extent to which they are managed well in a given work setting.

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Profit, MD, MPH, Principal Investigator — Stanford University; J. Bryan Sexton, PhD, Principal Investigator — Duke University
Locations (9):
- United States (9):
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Stanford University Medical Center, Stanford, California
  - Beth Israel Deconness Medical Center, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - University of North Carolina at Chapel Hill Children's Hospital, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas, Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
only research team will be accessing the data.

REFERENCES:
- [Background] Dyrbye LN, Shanafelt TD. Physician burnout: a potential threat to successful health care reform. JAMA. 2011 May 18;305(19):2009-10. doi: 10.1001/jama.2011.652. No abstract available. PMID 21586718
- [Background] Aiken LH, Sermeus W, Van den Heede K, Sloane DM, Busse R, McKee M, Bruyneel L, Rafferty AM, Griffiths P, Moreno-Casbas MT, Tishelman C, Scott A, Brzostek T, Kinnunen J, Schwendimann R, Heinen M, Zikos D, Sjetne IS, Smith HL, Kutney-Lee A. Patient safety, satisfaction, and quality of hospital care: cross sectional surveys of nurses and patients in 12 countries in Europe and the United States. BMJ. 2012 Mar 20;344:e1717. doi: 10.1136/bmj.e1717. PMID 22434089
- [Background] West CP, Tan AD, Shanafelt TD. Association of resident fatigue and distress with occupational blood and body fluid exposures and motor vehicle incidents. Mayo Clin Proc. 2012 Dec;87(12):1138-44. doi: 10.1016/j.mayocp.2012.07.021. PMID 23218084
- [Background] Fahrenkopf AM, Sectish TC, Barger LK, Sharek PJ, Lewin D, Chiang VW, Edwards S, Wiedermann BL, Landrigan CP. Rates of medication errors among depressed and burnt out residents: prospective cohort study. BMJ. 2008 Mar 1;336(7642):488-91. doi: 10.1136/bmj.39469.763218.BE. Epub 2008 Feb 7. PMID 18258931
- [Background] Sexton JB, Helmreich RL, Neilands TB, Rowan K, Vella K, Boyden J, Roberts PR, Thomas EJ. The Safety Attitudes Questionnaire: psychometric properties, benchmarking data, and emerging research. BMC Health Serv Res. 2006 Apr 3;6:44. doi: 10.1186/1472-6963-6-44. PMID 16584553
- [Background] Profit J, Sharek PJ, Amspoker AB, Kowalkowski MA, Nisbet CC, Thomas EJ, Chadwick WA, Sexton JB. Burnout in the NICU setting and its relation to safety culture. BMJ Qual Saf. 2014 Oct;23(10):806-13. doi: 10.1136/bmjqs-2014-002831. Epub 2014 Apr 17. PMID 24742780
- [Background] Sexton JB, Sharek PJ, Thomas EJ, Gould JB, Nisbet CC, Amspoker AB, Kowalkowski MA, Schwendimann R, Profit J. Exposure to Leadership WalkRounds in neonatal intensive care units is associated with a better patient safety culture and less caregiver burnout. BMJ Qual Saf. 2014 Oct;23(10):814-22. doi: 10.1136/bmjqs-2013-002042. Epub 2014 May 13. PMID 24825895
- [Background] van Wyk BE, Pillay-Van Wyk V. Preventive staff-support interventions for health workers. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD003541. doi: 10.1002/14651858.CD003541.pub2. PMID 20238322
- [Background] Sexton JB, Chadwick WA, Weiss KJ, Clarke A, Gould JB, Profit J. Assessing and Improving Health Care Worker Resilience in the NICU. E-PAS 2013:4150.7
- [Background] Ungar M. Researching and theorizing resilience across cultures and contexts. Prev Med. 2012 Nov;55(5):387-9. doi: 10.1016/j.ypmed.2012.07.021. Epub 2012 Aug 1. No abstract available. PMID 22884666
- [Background] Maslach C, Jackson SE. Maslach Burnout Inventory. Palo Alto, CA: Consulting Psychologists Press, Inc.; 1981
- [Background] Profit J, Gould JB, Zupancic JA, Stark AR, Wall KM, Kowalkowski MA, Mei M, Pietz K, Thomas EJ, Petersen LA. Formal selection of measures for a composite index of NICU quality of care: Baby-MONITOR. J Perinatol. 2011 Nov;31(11):702-10. doi: 10.1038/jp.2011.12. Epub 2011 Feb 24. PMID 21350429
- [Background] Ahola K, Vaananen A, Koskinen A, Kouvonen A, Shirom A. Burnout as a predictor of all-cause mortality among industrial employees: a 10-year prospective register-linkage study. J Psychosom Res. 2010 Jul;69(1):51-7. doi: 10.1016/j.jpsychores.2010.01.002. Epub 2010 Mar 19. PMID 20630263
- [Background] Kitaoka-Higashiguchi K, Morikawa Y, Miura K, Sakurai M, Ishizaki M, Kido T, Naruse Y, Nakagawa H. Burnout and risk factors for arteriosclerotic disease: follow-up study. J Occup Health. 2009;51(2):123-31. doi: 10.1539/joh.l8104. Epub 2009 Feb 10. PMID 19212087
- [Background] Guest RS, Baser R, Li Y, Scardino PT, Brown AE, Kissane DW. Cancer surgeons' distress and well-being, II: modifiable factors and the potential for organizational interventions. Ann Surg Oncol. 2011 May;18(5):1236-42. doi: 10.1245/s10434-011-1623-5. Epub 2011 Mar 12. PMID 21399883
- [Background] Campbell DA Jr, Sonnad SS, Eckhauser FE, Campbell KK, Greenfield LJ. Burnout among American surgeons. Surgery. 2001 Oct;130(4):696-702; discussion 702-5. doi: 10.1067/msy.2001.116676. PMID 11602901
- [Background] Geurts S, Rutte C, Peeters M. Antecedents and consequences of work-home interference among medical residents. Soc Sci Med. 1999 May;48(9):1135-48. doi: 10.1016/s0277-9536(98)00425-0. PMID 10220015
- [Background] Mealer M, Burnham EL, Goode CJ, Rothbaum B, Moss M. The prevalence and impact of post traumatic stress disorder and burnout syndrome in nurses. Depress Anxiety. 2009;26(12):1118-26. doi: 10.1002/da.20631. PMID 19918928
- [Background] Demir Zencirci A, Arslan S. Morning-evening type and burnout level as factors influencing sleep quality of shift nurses: a questionnaire study. Croat Med J. 2011 Aug 15;52(4):527-37. doi: 10.3325/cmj.2011.52.527. PMID 21853548
- [Background] Zhang Y, Feng X. The relationship between job satisfaction, burnout, and turnover intention among physicians from urban state-owned medical institutions in Hubei, China: a cross-sectional study. BMC Health Serv Res. 2011 Sep 24;11:235. doi: 10.1186/1472-6963-11-235. PMID 21943042
- [Background] Shelledy DC, Mikles SP, May DF, Youtsey JW. Analysis of job satisfaction, burnout, and intent of respiratory care practitioners to leave the field or the job. Respir Care. 1992 Jan;37(1):46-60. PMID 10145581
- [Background] Shanafelt TD, Bradley KA, Wipf JE, Back AL. Burnout and self-reported patient care in an internal medicine residency program. Ann Intern Med. 2002 Mar 5;136(5):358-67. doi: 10.7326/0003-4819-136-5-200203050-00008. PMID 11874308
- [Background] Meeusen VC, Van Dam K, Brown-Mahoney C, Van Zundert AA, Knape HT. Understanding nurse anesthetists' intention to leave their job: how burnout and job satisfaction mediate the impact of personality and workplace characteristics. Health Care Manage Rev. 2011 Apr-Jun;36(2):155-63. doi: 10.1097/HMR.0b013e3181fb0f41. PMID 21317664
- [Background] McMurray JE, Linzer M, Konrad TR, Douglas J, Shugerman R, Nelson K. The work lives of women physicians results from the physician work life study. The SGIM Career Satisfaction Study Group. J Gen Intern Med. 2000 Jun;15(6):372-80. doi: 10.1111/j.1525-1497.2000.im9908009.x. PMID 10886471
- [Background] West CP, Huschka MM, Novotny PJ, Sloan JA, Kolars JC, Habermann TM, Shanafelt TD. Association of perceived medical errors with resident distress and empathy: a prospective longitudinal study. JAMA. 2006 Sep 6;296(9):1071-8. doi: 10.1001/jama.296.9.1071. PMID 16954486
- [Background] Shanafelt TD, Balch CM, Bechamps G, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag J. Burnout and medical errors among American surgeons. Ann Surg. 2010 Jun;251(6):995-1000. doi: 10.1097/SLA.0b013e3181bfdab3. PMID 19934755
- [Background] Prins JT, van der Heijden FM, Hoekstra-Weebers JE, Bakker AB, van de Wiel HB, Jacobs B, Gazendam-Donofrio SM. Burnout, engagement and resident physicians' self-reported errors. Psychol Health Med. 2009 Dec;14(6):654-66. doi: 10.1080/13548500903311554. PMID 20183538
- [Background] Rochefort CM, Clarke SP. Nurses' work environments, care rationing, job outcomes, and quality of care on neonatal units. J Adv Nurs. 2010 Oct;66(10):2213-24. doi: 10.1111/j.1365-2648.2010.05376.x. Epub 2010 Jul 2. PMID 20626479
- [Background] Aiken LH, Clarke SP, Sloane DM, Sochalski J, Silber JH. Hospital nurse staffing and patient mortality, nurse burnout, and job dissatisfaction. JAMA. 2002 Oct 23-30;288(16):1987-93. doi: 10.1001/jama.288.16.1987. PMID 12387650
- [Background] Cherniss C. Staff Burnout: Job Stress in the Human Services. Beverly Hills, CA: Sage Publications; 1980
- [Background] Bellieni CV, Righetti P, Ciampa R, Iacoponi F, Coviello C, Buonocore G. Assessing burnout among neonatologists. J Matern Fetal Neonatal Med. 2012 Oct;25(10):2130-4. doi: 10.3109/14767058.2012.666590. Epub 2012 May 10. PMID 22571319
- [Background] Shanafelt TD, Balch CM, Bechamps GJ, Russell T, Dyrbye L, Satele D, Collicott P, Novotny PJ, Sloan J, Freischlag JA. Burnout and career satisfaction among American surgeons. Ann Surg. 2009 Sep;250(3):463-71. doi: 10.1097/SLA.0b013e3181ac4dfd. PMID 19730177
- [Background] Cimiotti JP, Aiken LH, Sloane DM, Wu ES. Nurse staffing, burnout, and health care-associated infection. Am J Infect Control. 2012 Aug;40(6):486-90. doi: 10.1016/j.ajic.2012.02.029. PMID 22854376
- [Background] Sexton JB, Berenholtz SM, Goeschel CA, Watson SR, Holzmueller CG, Thompson DA, Hyzy RC, Marsteller JA, Schumacher K, Pronovost PJ. Assessing and improving safety climate in a large cohort of intensive care units. Crit Care Med. 2011 May;39(5):934-9. doi: 10.1097/CCM.0b013e318206d26c. PMID 21297460
- [Background] Marsteller JA, Sexton JB, Hsu YJ, Hsiao CJ, Holzmueller CG, Pronovost PJ, Thompson DA. A multicenter, phased, cluster-randomized controlled trial to reduce central line-associated bloodstream infections in intensive care units*. Crit Care Med. 2012 Nov;40(11):2933-9. doi: 10.1097/CCM.0b013e31825fd4d8. PMID 22890251
- [Background] Marshall RE, Kasman C. Burnout in the neonatal intensive care unit. Pediatrics. 1980 Jun;65(6):1161-5. PMID 7375242
- [Background] Krasner MS, Epstein RM, Beckman H, Suchman AL, Chapman B, Mooney CJ, Quill TE. Association of an educational program in mindful communication with burnout, empathy, and attitudes among primary care physicians. JAMA. 2009 Sep 23;302(12):1284-93. doi: 10.1001/jama.2009.1384. PMID 19773563
- [Background] McCray LW, Cronholm PF, Bogner HR, Gallo JJ, Neill RA. Resident physician burnout: is there hope? Fam Med. 2008 Oct;40(9):626-32. PMID 18830837
- [Background] Rowe MM. Teaching health-care providers coping: results of a two-year study. J Behav Med. 1999 Oct;22(5):511-27. doi: 10.1023/a:1018661508593. PMID 10586384
- [Background] West CP, Dyrbye LN, Rabatin JT, Call TG, Davidson JH, Multari A, Romanski SA, Hellyer JM, Sloan JA, Shanafelt TD. Intervention to promote physician well-being, job satisfaction, and professionalism: a randomized clinical trial. JAMA Intern Med. 2014 Apr;174(4):527-33. doi: 10.1001/jamainternmed.2013.14387. PMID 24515493
- [Background] Sin NL, Lyubomirsky S. Enhancing well-being and alleviating depressive symptoms with positive psychology interventions: a practice-friendly meta-analysis. J Clin Psychol. 2009 May;65(5):467-87. doi: 10.1002/jclp.20593. PMID 19301241
- [Background] Pronovost P, Needham D, Berenholtz S, Sinopoli D, Chu H, Cosgrove S, Sexton B, Hyzy R, Welsh R, Roth G, Bander J, Kepros J, Goeschel C. An intervention to decrease catheter-related bloodstream infections in the ICU. N Engl J Med. 2006 Dec 28;355(26):2725-32. doi: 10.1056/NEJMoa061115. PMID 17192537
- [Background] Cohen S, Wills TA. Stress, social support, and the buffering hypothesis. Psychol Bull. 1985 Sep;98(2):310-57. No abstract available. PMID 3901065
- [Background] Brown C, Hofer T, Johal A, Thomson R, Nicholl J, Franklin BD, Lilford RJ. An epistemology of patient safety research: a framework for study design and interpretation. Part 2. Study design. Qual Saf Health Care. 2008 Jun;17(3):163-9. doi: 10.1136/qshc.2007.023648. PMID 18519621
- [Background] Hussey MA, Hughes JP. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. 2007 Feb;28(2):182-91. doi: 10.1016/j.cct.2006.05.007. Epub 2006 Jul 7. PMID 16829207
- [Background] Kao LS, Lew DF, Doyle PD, Carrick MM, Jordan VS, Thomas EJ, Lally KP. A tale of 2 hospitals: a staggered cohort study of targeted interventions to improve compliance with antibiotic prophylaxis guidelines. Surgery. 2010 Aug;148(2):255-62. doi: 10.1016/j.surg.2010.04.003. Epub 2010 May 21. PMID 20494387
- [Background] Profit J, Zupancic JA, Gould JB, Pietz K, Kowalkowski MA, Draper D, Hysong SJ, Petersen LA. Correlation of neonatal intensive care unit performance across multiple measures of quality of care. JAMA Pediatr. 2013 Jan;167(1):47-54. doi: 10.1001/jamapediatrics.2013.418. PMID 23403539
- [Background] Profit J, Kowalkowski MA, Zupancic JA, Pietz K, Richardson P, Draper D, Hysong SJ, Thomas EJ, Petersen LA, Gould JB. Baby-MONITOR: a composite indicator of NICU quality. Pediatrics. 2014 Jul;134(1):74-82. doi: 10.1542/peds.2013-3552. Epub 2014 Jun 2. PMID 24918221
- [Background] Jarvis P. Adult Education and Lifelong Learning: Theory and Practice. 4th ed. New York, NY: Routledge; 2010
- [Background] Profit J, Etchegaray J, Petersen LA, Sexton JB, Hysong SJ, Mei M, Thomas EJ. Neonatal intensive care unit safety culture varies widely. Arch Dis Child Fetal Neonatal Ed. 2012 Mar;97(2):F120-6. doi: 10.1136/archdischild-2011-300635. Epub 2011 Sep 19. PMID 21930691
- [Background] Edwards D, Burnard P, Coyle D, Fothergill A, Hannigan B. A stepwise multivariate analysis of factors that contribute to stress for mental health nurses working in the community. J Adv Nurs. 2001 Dec;36(6):805-13. doi: 10.1046/j.1365-2648.2001.02035.x. PMID 11903710
- [Background] Kohout FJ, Berkman LF, Evans DA, Cornoni-Huntley J. Two shorter forms of the CES-D (Center for Epidemiological Studies Depression) depression symptoms index. J Aging Health. 1993 May;5(2):179-93. doi: 10.1177/089826439300500202. PMID 10125443
- [Background] Pennebaker JW, Colder M, Sharp LK. Accelerating the coping process. J Pers Soc Psychol. 1990 Mar;58(3):528-537. doi: 10.1037//0022-3514.58.3.528. PMID 2324942
- [Background] Vogus TJ, Sutcliffe KM. The impact of safety organizing, trusted leadership, and care pathways on reported medication errors in hospital nursing units. Med Care. 2007 Oct;45(10):997-1002. doi: 10.1097/MLR.0b013e318053674f. PMID 17890998
- [Background] Profit J, Etchegaray J, Petersen LA, Sexton JB, Hysong SJ, Mei M, Thomas EJ. The Safety Attitudes Questionnaire as a tool for benchmarking safety culture in the NICU. Arch Dis Child Fetal Neonatal Ed. 2012 Mar;97(2):F127-32. doi: 10.1136/archdischild-2011-300612. PMID 22337935
- [Background] Profit J, Weiss K, Clarke A, Gest AL, Sexton JB. NICU Caregiver Burnout, Happiness, and Three Good Things. Pediatric Academic Societies' Annual Meeting 2014;E-PAS 3844.652
- [Background] Maslach C, Jackson S. The measurement of experienced burnout. J Occ Behav 1981;2:99-113
- [Background] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Background] Shanafelt TD, West CP, Sloan JA, Novotny PJ, Poland GA, Menaker R, Rummans TA, Dyrbye LN. Career fit and burnout among academic faculty. Arch Intern Med. 2009 May 25;169(10):990-5. doi: 10.1001/archinternmed.2009.70. PMID 19468093
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Lyubomirsky S, Ross L. Changes in attractiveness of elected, rejected, and precluded alternatives: a comparison of happy and unhappy individuals. J Pers Soc Psychol. 1999 Jun;76(6):988-1007. doi: 10.1037//0022-3514.76.6.988. PMID 10402682
- [Background] Howell RT, Rodzon KS, Kurai M, Sanchez AH. A validation of well-being and happiness surveys for administration via the Internet. Behav Res Methods. 2010 Aug;42(3):775-84. doi: 10.3758/BRM.42.3.775. PMID 20805600
- [Background] Hudson DW, Berenholtz SM, Thomas EJ, Sexton BJ. A safety culture primer for the critical care clinician: the role of culture in patient safety and quality improvement. Contemp Crit Care 2009;7:1-12
- [Background] Pronovost P, Weast B. Implementing and validating a comprehensive unit-based safety program. J Patient Saf 2005:33-40
- [Background] Pettker CM, Thung SF, Norwitz ER, Buhimschi CS, Raab CA, Copel JA, Kuczynski E, Lockwood CJ, Funai EF. Impact of a comprehensive patient safety strategy on obstetric adverse events. Am J Obstet Gynecol. 2009 May;200(5):492.e1-8. doi: 10.1016/j.ajog.2009.01.022. Epub 2009 Feb 27. PMID 19249729
- [Background] Wolf FA, Way LW, Stewart L. The efficacy of medical team training: improved team performance and decreased operating room delays: a detailed analysis of 4863 cases. Ann Surg. 2010 Sep;252(3):477-83; discussion 483-5. doi: 10.1097/SLA.0b013e3181f1c091. PMID 20739848
- [Background] Pronovost PJ, Berenholtz SM, Goeschel C, Thom I, Watson SR, Holzmueller CG, Lyon JS, Lubomski LH, Thompson DA, Needham D, Hyzy R, Welsh R, Roth G, Bander J, Morlock L, Sexton JB. Improving patient safety in intensive care units in Michigan. J Crit Care. 2008 Jun;23(2):207-21. doi: 10.1016/j.jcrc.2007.09.002. PMID 18538214
- [Background] Profit J, Sexton JB, Thomas EJ, et al. Higher Safety Culture among Neonatal Intensive Care Units That Participate in Quality Improvement Collaboratives. E-PAS 2012:2920.350
- [Background] Profit J, Lee HC, Sharek PJ, et al. NICU Safety Culture: The Effect of Choice of Instrument on Benchmarking. Pediatrics 2014;Under review
- [Background] Profit J, Typpo KV, Hysong SJ, Woodard LD, Kallen MA, Petersen LA. Improving benchmarking by using an explicit framework for the development of composite indicators: an example using pediatric quality of care. Implement Sci. 2010 Feb 9;5:13. doi: 10.1186/1748-5908-5-13. PMID 20181129
- [Background] Sexton JB, Sharek PJ, Gould JB, et al. Prevalence of Emotional Exhaustion in a Cohort of 21 Neonatal Intensive Care Units. E-PAS 2012:2920.351
- [Background] Profit J, Sharek PJ, Thomas EJ, et al. Clinical Outcomes among VLBW Infants and the Links to Subsequent Perceptions of NICU Safety Culture. E-PAS 2013:2922.356
- [Background] Chadwick WA, Fullwood C, Mullin L, Browning B, Schifer C, Pietrusik J. Webinar Implementation for the Science of Enhancing Resilience (WISER): the development and evaluation of WISER 1.0. Duke University Medical School Research Day. Durham, NC2012
- [Background] Timmel J, Kent PS, Holzmueller CG, Paine L, Schulick RD, Pronovost PJ. Impact of the Comprehensive Unit-based Safety Program (CUSP) on safety culture in a surgical inpatient unit. Jt Comm J Qual Patient Saf. 2010 Jun;36(6):252-60. doi: 10.1016/s1553-7250(10)36040-5. PMID 20564886
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Emmons RA, McCullough ME. Counting blessings versus burdens: an experimental investigation of gratitude and subjective well-being in daily life. J Pers Soc Psychol. 2003 Feb;84(2):377-89. doi: 10.1037//0022-3514.84.2.377. PMID 12585811
- [Result] Profit J, Adair KC, Cui X, Mitchell B, Brandon D, Tawfik DS, Rigdon J, Gould JB, Lee HC, Timpson WL, McCaffrey MJ, Davis AS, Pammi M, Matthews M, Stark AR, Papile LA, Thomas E, Cotten M, Khan A, Sexton JB. Randomized controlled trial of the "WISER" intervention to reduce healthcare worker burnout. J Perinatol. 2021 Sep;41(9):2225-2234. doi: 10.1038/s41372-021-01100-y. Epub 2021 Aug 9. PMID 34366432
- [Derived] Profit J, Cui X, Tawfik D, Adair KC, Sexton JB. "WISER" intervention to reduce healthcare worker burnout - 1 year follow up. J Perinatol. 2024 Dec;44(12):1719-1723. doi: 10.1038/s41372-024-01993-5. Epub 2024 May 11. PMID 38734802
- [Derived] Sexton JB, Adair KC, Cui X, Tawfik DS, Profit J. Effectiveness of a bite-sized web-based intervention to improve healthcare worker wellbeing: A randomized clinical trial of WISER. Front Public Health. 2022 Dec 8;10:1016407. doi: 10.3389/fpubh.2022.1016407. eCollection 2022. PMID 36568789
- [Derived] Kunzler AM, Helmreich I, Chmitorz A, Konig J, Binder H, Wessa M, Lieb K. Psychological interventions to foster resilience in healthcare professionals. Cochrane Database Syst Rev. 2020 Jul 5;7(7):CD012527. doi: 10.1002/14651858.CD012527.pub2. PMID 32627860